CLINICAL TRIAL: NCT01527383
Title: A Phase II Randomized, Placebo-Controlled Clinical Trial to Study the Safety and Immunogenicity of V212 in Adult Patients With Autoimmune Disease
Brief Title: A Study to Evaluate the Safety and Immunogenicity of Inactivated Varicella Zoster Virus (VZV) Vaccine in Adults With Autoimmune Disease (V212-009)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: V212-009; V212-009 (Other: Merck Protocol Number); 2011-002313-11 (EudraCT Number)
Record Dates: First submitted 2012-01-16; First posted 2012-02-07 (Estimated); Results first posted 2019-01-14 (Actual); Last update posted 2019-01-14 (Actual); Status verified 2019-01

CONDITIONS: Herpes Zoster
Keywords: Shingles
MeSH Terms: conditions — Herpes Zoster | interventions — Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- V212 (Experimental): Participants receive V212 as a 0.5 mL subcutaneous injection in a four-dose regimen, approximately 30 days apart, preferably in the deltoid area of the arm, alternating arms for each dose.
  Interventions: Biological: V212
- Placebo (Placebo Comparator): Participants receive placebo as a 0.5 mL subcutaneous injection in a four-dose regimen, approximately 30 days apart, preferably in the deltoid area of the arm, alternating arms for each dose.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: V212 — V212 viral antigen for HZ
  Other Names: Inactivated Varicella-Zoster (VZV) vaccine
  Arms: V212
Biological: Placebo — Placebo comparator to V212 vaccine
  Arms: Placebo

SUMMARY:
This is a study to evaluate the safety and immunogenicity of V212 vaccine in adults with autoimmune disease, including participants with rheumatoid arthritis, psoriatic arthritis, psoriasis, inflammatory bowel disease, systemic lupus erythematosus, multiple sclerosis, and other similar diseases. The primary hypothesis is that vaccination with V212 vaccine will elicit significant VZV-specific immune responses at approximately 28 days after vaccination 4. The statistical criterion for significance requires that the lower bound of the 2-sided 95% confidence interval of the geometric mean fold rise in vaccine recipients is >1.0.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with an autoimmune disease
* Clinically stable disease for at least 30 days before enrollment
* Not likely to undergo hematopoietic stem cell transplantation during the study period
* Receiving at least one parenteral or oral biologic agent, such as a Tumor Necrosis factor (TNF) alpha inhibitor, or a parenteral or oral non-biologic therapy, at a stable dose for at least 3 months, with no planned or anticipated changes
* History of varicella, antibodies to VZV, or residence for at least 30 years in a country with endemic VZV infection, or if participant is less than 30 years old, attended primary or secondary school in a country with endemic VZV infection

Exclusion Criteria:

* Prior history of Herpes Zoster (shingles) within 1 year before enrollment
* Prior varicella or zoster vaccine
* Active central nervous system lupus erythematosus requiring therapeutic intervention within 90 days of enrollment
* Prior or planned therapy containing rituximab or other anti-Cluster of Differentiation (CD) 20 monoclonal antibodies from 3 months before enrollment through 28 days postdose 4
* Systemic corticosteroid therapy, prednisone, or equivalent over 40 mg daily at the time of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 354 (Actual)
Dates: Start 2012-02-21 (Actual); Primary Completion 2013-02-26 (Actual); Study Completion 2013-02-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Eberhardson M, Hall S, Papp KA, Sterling TM, Stek JE, Pang L, Zhao Y, Parrino J, Popmihajlov Z. Safety and Immunogenicity of Inactivated Varicella-Zoster Virus Vaccine in Adults With Autoimmune Disease: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Clinical Trial. Clin Infect Dis. 2017 Oct 1;65(7):1174-1182. doi: 10.1093/cid/cix484. PMID 29126292

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 362 participants were screened and 354 were enrolled.
Groups:
- V212: Participants received V212 as a 0.5 mL subcutaneous injection in a four-dose regimen, approximately 30 days apart, preferably in the deltoid area of the arm, alternating arms for each dose.
- Placebo: Participants received placebo as a 0.5 mL subcutaneous injection in a four-dose regimen, approximately 30 days apart, preferably in the deltoid area of the arm, alternating arms for each dose.
Period: Overall Study
Arm/Group | V212 | Placebo
Started | 292 | 62
Vaccination 1 (Day 1) | 291 | 62
Vaccination 2 (~Day 30) | 283 | 61
Vaccination 3 (~Day 60) | 278 | 58
Vaccination 4 (~Day 90) | 277 | 58
Completed | 277 | 58
Not Completed | 15 | 4
Not completed — Adverse Event | 5 | 0
Not completed — Lost to Follow-up | 3 | 0
Not completed — Physician Decision | 2 | 0
Not completed — Pregnancy | 1 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Screen failure | 1 | 0
Not completed — Participant moved | 0 | 1
Not completed — Withdrawal by Subject | 2 | 3

BASELINE CHARACTERISTICS:
Population: All enrolled participants
Groups:
- Total: Total of all reporting groups
Arm/Group | V212 | Placebo | Total
Number analyzed (Participants) | 292 | 62 | 354
Age, Customized [Number; unit: Participants]
  18 to 49 years | 118 | 27 | 145
  50 to 59 years | 89 | 14 | 103
  60 to 69 years | 65 | 12 | 77
  70 to 79 years | 20 | 6 | 26
  80+ years | 0 | 3 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 189 | 37 | 226
  Male | 103 | 25 | 128
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 43 | 9 | 52
  Not Hispanic or Latino | 248 | 53 | 301
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 23 | 5 | 28
  White | 239 | 49 | 288
  More than one race | 26 | 8 | 34
  Unknown or Not Reported | 0 | 0 | 0
Autoimmune Therapy Regimen: Biologic or Non-biologic [Count of Participants; unit: Participants]
  Biologic autoimmune therapy regimen | 142 | 28 | 170
  Non-biologic autoimmune therapy regimen | 150 | 34 | 184

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Fold Rise (GMFR) in Varicella-Zoster (VZV) Antibody Responses Measured by Glycoprotein Enzyme-linked Immunosorbent Assay (gpELISA)
Description: Serum samples were tested for antibody response using a gpELISA. The GMFR is response at approximately 28 days postdose 4 / response predose on Day 1.
Time Frame: Baseline and ~28 days after Vaccination 4 (~Day 118)
Population: Participants with Day 1 and/or postdose data available. This outcome measure applied only to participants who received V212; placebo participants were not assessed for this outcome.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | V212
Number analyzed (Participants) | 176
Ratio | 1.57 [1.44 to 1.72]
Statistical Analysis 1: Comparison: V212; Test type: Other; p < 0.0001, Longitudinal regression; Visit and stratification factor (biologic or non-biologic autoimmune therapy) were covariates; The statistical criterion for significance requires that the lower bound of the 2-sided 95% confidence interval of the geometric mean fold rise in vaccine recipients is >1.0

2. Primary Outcome: GMFR in VZV Antibody Response Measured by VZV Interferon-gamma (IFN-g) Enzyme-linked Immunospot (ELISPOT) Assay
Description: Serum samples were tested for activity using a VZV ELISPOT assay. The assay detects IFN-γ-secreting, VZV-specific cells from peripheral blood mononuclear cells (PBMCs). The unit of measure of the assay is ELISPOT cell count / 10^6 PBMCs, and is expressed as geometric mean count (GMC). The GMFR is GMC at ~28 days after Vaccination 4 / GMC predose on Day 1.
Time Frame: Baseline and ~28 days after Vaccination 4 (~Day 118)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | V212
Number analyzed (Participants) | 176
Ratio | 2.01 [1.57 to 2.58]
Statistical Analysis 1: Comparison: V212; Test type: Other; p < 0.0001, Longitudinal regression; Visit and stratification factor (biologic or non-biologic autoimmune therapy) were covariates; [other analysis details as in outcome 1, analysis 1]

3. Primary Outcome: Percentage of Participants With a Serious Adverse Event
Description: A serious adverse event (SAE) is defined as an adverse event that resulted in death, was life threatening, resulted in persistent or significant disability or incapacity, resulted in or prolonged a hospitalization, is a congenital anomaly or birth defect, is a cancer, was an overdose, or was an important medical event based on appropriate medical judgment. The percentage of participants with one or more SAE was assessed.
Time Frame: Up to ~28 days after Vaccination 4 (~Day 118)
Population: All participants who received at least one dose of vaccine and had safety follow-up
Measure: Number; unit: Percentage of participants
Arm/Group | V212 | Placebo
Number analyzed (Participants) | 289 | 62
Percentage of participants | 2.8 | 1.6

4. Secondary Outcome: Percentage of Participants With an Injection-site Adverse Event Prompted on the Vaccination Report Card
Description: An adverse event (AE) is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study vaccine, whether or not considered related to the use of the study vaccine. Any worsening of a preexisting condition which is temporally associated with the use of the study vaccine is also an AE. Vaccination Report Card (VRC)-prompted injection-site AEs were erythema, pain, and swelling. The percentage of participants with one or more VRC-prompted injection-site AE was assessed.
Time Frame: Up to Day 5 after any vaccination
Population: All participants who received at least one dose of vaccine and had safety follow-up
Measure: Number; unit: Percentage of participants
Arm/Group | V212 | Placebo
Number analyzed (Participants) | 289 | 62
Percentage of participants
  Injection-site erythema | 46.0 | 1.6
  Injection-site pain | 42.2 | 14.5
  Injection-site swelling | 40.1 | 4.8

5. Secondary Outcome: Percentage of Participants With a Systemic Adverse Event Prompted on the Vaccination Report Card
Description: An AE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study vaccine, whether or not considered related to the use of the study vaccine. Any worsening of a preexisting condition which is temporally associated with the use of the study vaccine is also an AE. VRC-prompted systemic AEs included non-injection-site varicella-like and HZ-like rashes. The percentage of participants with one or more VRC-prompted systemic AE was assessed.
Time Frame: Up to ~28 days after Vaccination 4 (~Day 118)
Population: All participants who received at least one dose of vaccine and had safety follow-up
Measure: Number; unit: Percentage of participants
Arm/Group | V212 | Placebo
Number analyzed (Participants) | 289 | 62
Percentage of participants | 51.6 | 46.8

6. Secondary Outcome: Percentage of Participants With Elevated Temperature Prompted on the Vaccination Report Card
Description: Elevated temperature is defined as ≥100.4 °F (≥38.0 °C), oral equivalent. The percentage of participants with VRC-prompted elevated temperature was assessed.
Time Frame: Up to ~28 days after Vaccination 4 (~Day 118)
Population: All participants who received at least one dose of vaccine and had safety follow-up
Measure: Number; unit: Percentage of participants
Arm/Group | V212 | Placebo
Number analyzed (Participants) | 284 | 61
Percentage of participants | 7.0 | 4.9

ADVERSE EVENTS:
Time Frame: Up to Day 140
Description: All participants who received at least one dose of vaccine and had safety follow-up
Arm/Group | V212 | Placebo
All-Cause Mortality (participants affected / at risk) | 1/289 | 0/62
Serious Adverse Events (participants affected / at risk) | 9/289 | 1/62
Other Adverse Events (participants affected / at risk) | 171/289 | 11/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V212 (N=289) | Placebo (N=62)
Anaemia haemolytic autoimmune (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Keratitis (Eye disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Amnesia (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V212 (N=289) | Placebo (N=62)
Injection site erythema (General disorders) | 133 (318) | 1 (1)
Injection site pain (General disorders) | 122 (270) | 9 (11)
Injection site pruritus (General disorders) | 24 (44) | 0 (0)
Injection site swelling (General disorders) | 116 (255) | 3 (3)
Nasopharyngitis (Infections and infestations) | 17 (19) | 1 (1)
Headache (Nervous system disorders) | 21 (30) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission.